CLINICAL TRIAL: NCT02772575
Title: A PILOT STUDY TO IDENTIFY MOLECULAR PREDICTORS OF SENSITIVITY AND RESISTANCE TO TRANS-ARTERIAL EMBOLIZATION OF PRIMARY LIVER TUMORS AND LIVER METASTASES
Brief Title: A Study to See if we Can Predict How Your Liver Tumor or Liver Metastases Will Respond to Trans-Arterial Embolization (TAE)
Status: Withdrawn | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-385
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Liver Cancer; Liver Metastases
Keywords: MOLECULAR PREDICTORS; Hepatic trans-arterial embolization (TAE); 16-385
MeSH Terms: conditions — Liver Neoplasms | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue blood

GROUPS / COHORTS (1):
- patients with primary liver or liver metastases: A biopsy will be performed as standard of care either at time of Hepatic trans-arterial embolization (TAE) or within 4 months prior to TAE. TAE is a standard of care procedure. Within 8 weeks of TAE, patient will have a clinic visit which will include medical history, physical examination, vital signs, EKG (if one is not available), and ECOG assessment. Additionally a dedicated liver CT or MR will be obtained as well as standard of care labs. IMPACT blood test will be performed at the time of any of the standard of care labs. As IMPACT platform at MSKCC continually evolves to include more genes, we will use the platform available at the time of initiation of the protocol, therefore all patients will be subjected to the same platform. RNA-seq has been demonstrated to be superior in detecting low abundance transcripts, demonstrating a broader dynamic range, and detecting different isoforms and genetic variants.
  Interventions: Procedure: Hepatic trans-arterial embolization (TAE); Device: MRI/CT scan; Procedure: biopsy; Other: blood draw

INTERVENTIONS:
Procedure: Hepatic trans-arterial embolization (TAE)
Device: MRI/CT scan
Procedure: biopsy
Other: blood draw

SUMMARY:
The purpose of this study is to see if certain genes the tumor can help predict how the tumor will respond to Trans-Arterial Embolization (TAE). A gene is the basic physical and functional unit of heredity. Genes are made up of DNA; DNA (deoxyribonucleic acid) is the hereditary material in humans. Identifying a gene that can predict how liver tumors will respond to TAE will also help to determine if adjuvant therapy will be needed after TAE.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic evidence of primary liver cancer or liver metastases
* Indication of TAE for the treatment of liver tumor
* Age ≥ 18 years
* Available tissue with adequate tissue for analysis, verified by a pathologist

Exclusion Criteria:

* History of a second active malignancy with evidence of metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, listed protocol investigators, or Interventional Radiology research team at Memorial Sloan Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
response | within 4 weeks
  Response will be categorized using standard mRECIST criteria. Tumor response will be catalogued as follows:
  Complete Response (CR): Disappearance of any intratumoral arterial enhancement in all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions.
  Stable Disease (SD): Any cases that do not qualify for either partial response or progressive disease. Progressive Disease (PD): An increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the of viable (enhancing) target lesions recorded since treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Etay Ziv, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/